CLINICAL TRIAL: NCT02790697
Title: Clinical Evaluation of the Ease of Use of a New Indirect Calorimeter for Energy Expenditure Measurement in ICU Patients: The ICALIC International Multicentric Study
Brief Title: The ICALIC Accuracy Validation in Geneva Study
Acronym: ICALIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Claude Pichard, Claude Pichard, MD, PhD, University Hospital, Geneva
Other Study IDs: 15-137_Addendum
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Critical Illness
Keywords: Indirect calorimetry; ICALIC Study; Energy expenditure; VO2; VCO2; Respiratory quotient
MeSH Terms: conditions — Critical Illness | interventions — Calorimetry, Indirect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically ventilated ICU patient: Indirect calorimetry measurements will be conducted using the new calorimeter and the mass spectrometer system at the same time for all enrolled patients.
  Interventions: Other: Indirect calorimetry

INTERVENTIONS:
Other: Indirect calorimetry — Indirect calorimetry will be conducted using the new calorimeter and mixing chamber method using the mass spectrometer.

SUMMARY:
This study aims at validating the accuracy of the new indirect calorimeter (Q-NRG, COSMED, Italy), developed for the ICALIC multicenter study. The validation of accuracy will only be conducted in Geneva center.

The measurements made with the new calorimeter will be compared to the measurements by the mixing chamber method using a mass spectrometer (MAX300-LG, Extrel, USA) for gas composition analysis.

DETAILED DESCRIPTION:
Indirect calorimetry is a method to measure energy expenditure of human subjects by analyzing patient breath gas to measure the amount (volume) of oxygen consumption (VO2) and CO2 production (VCO2). Energy expenditure is calculated by the Weir's equation using the measured VO2 and VCO2 values.

The new calorimeter is equipped with a disposable in-line pneumotach flowmeter, which measures the flow of exhaled gas of patients directly within the mechanical ventilator circuit. It also samples small amount of inhaled and exhaled gas to measure the inhaled and exhaled O2 and CO2 compositions. The new dynamic micro-mixing chamber technique is used to meaure VO2 and VCO2 to derive the energy expenditure.

The mass spectrometer measures the inhaled and exhaled gas compositions. The mass spectrometer samples inhaled gas from the mechanical ventilator circuit. A mixing chamber system is used to collect the expired gas from the outlet of the mechanical ventilator. The collected gas is measured for the second time after diluting with a constant flow of ambient air, which is monitored by an independent mass flow meter. The volume of the expired gas is calculated by comparison of the concentrations of exhaled gas before and after the dilution. The measurements will be used to calculate the VO2 and VCO2 to derive the energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

• Mechanically ventilated adult ICU patients

Exclusion Criteria:

* Fraction of inhaled oxygen (FIO2) > 70%
* Positive end expiratory pressure (PEEP) >10cmH2O
* Peak ventilatory pressure > 30cmH2O
* Presence of air leaks from thoracic drain tube
* Changes in vasoactive agent dose (>20%, <1 hr before and/or during IC)
* Agitation or change in sedative dose (>20%, <1 hr before and/or during IC)
* Change in body temperature (>0.5°C, <1 hr before and/or during IC)
* Expected duration of ICU stay < 24 hours
* Expected survival of the patient < 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated adult ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-09-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Energy expenditure | immediately after the measurement
  Energy expenditure calculated as a result of VO2 and VCO2 measurements

SECONDARY OUTCOMES:
Accuracy of VO2 | immediately after the measurement
  Volume of oxygen consumption
Accuracy of VCO2 | immediately after the measurement
  Volume of CO2 production
Respiratory quotient (RQ) | immediately after the measurement
  RQ calculated as a ratio of VCO2 to VO2

CONTACTS AND LOCATIONS:
Overall Officials: Claude Pichard, MD, PhD, Principal Investigator — Clinical Nutrition, Geneva University Hospital
Locations (1):
- Service of Intensive Care, Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No